CLINICAL TRIAL: NCT04897984
Title: The Kinetics of LEAP2 in Man
Brief Title: LEAP2 Kinetics in Healthy Individuals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, head of department, University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEAP2 kinetics
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The study is designed as a clinical study involving one experimental study day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver-enriched antimicrobial peptide 2 (Experimental): IV infusion of LEAP2, 2 hours
  Interventions: Biological: Liver-enriched antimicrobial peptide 2

INTERVENTIONS:
Biological: Liver-enriched antimicrobial peptide 2 — IV infusion of LEAP2, 2 hours

SUMMARY:
The study aims to investigate the kinetics of the naturally occurring peptide liver-enriched antimicrobial peptide 2 (LEAP-2) in healthy volunteers. The overall objective is to investigate the physiological importance of LEAP-2 in healthy subjects.

DETAILED DESCRIPTION:
In a recent study, the molecular phenotype of enteroendocrine cells in the small intestine before and after Roux-en-Y Gastric Bypass (RYGB) surgery in obese individuals was examined. Enteroendocrine cells were identified and isolated from intestinal biopsies and analysed for differentially expressed genes by Illumina High Throughput RNA-sequencing. It was discovered that the gene encoding liver-enriched antimicrobial peptide 2 (LEAP2), a naturally occurring peptide in humans, was significantly upregulated compared to baseline expression. Interestingly, LEAP2 was recently shown to antagonize ghrelin function in response to feeding in mice. Moreover, the mature murine LEAP2 peptide is identical in mice and humans. Thus, LEAP2 has been identified as an endogenous peptide that may be able to alter feeding behaviour and maintenance of glucose levels during calorie restriction.

This study aims to investigate the kinetics of exogenous LEAP2 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men
* Age between 18 and 25 years
* Body mass index between 20-35 kg/m2
* Informed consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary and/or gastrointestinal disorder(s)
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Allergy or intolerance to ingredients included in the standardised meals
* First-degree relatives with diabetes and/or glycated haemoglobin (HbA1c) >48 mmol/mol
* Regular tobacco smoking or use of other nicotine-containing products
* Any ongoing medication that the investigator evaluates would interfere with trial participation.
* Any physical or psychological condition that the investigator evaluates would interfere with trial participation including any acute or chronic illnesses

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of LEAP2 | -30 to 270 minutes
  Plasma concentrations of LEAP2

SECONDARY OUTCOMES:
VAS | -30 to 270 minutes
  Visual analogue scales (VASs) assessing appetite, satiety and hunger sensations (from 0 to 10 cm on a scale = from mimimum to maximum sensation)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No